CLINICAL TRIAL: NCT02373644
Title: Spinal Manipulation and Dry Needling Versus Conventional Physical Therapy in Patients With Sacroiliac Dysfunction: a Multi-center Randomized Clinical Trial
Brief Title: Spinal Manipulation and Dry Needling Versus Conventional Physical Therapy in Patients With Sacroiliac Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, DPT MSc FAAOMPT, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT0004
Record Dates: First submitted 2015-02-10; First posted 2015-02-27 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2019-10

CONDITIONS: Sacroiliac Joint Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HVLA Thrust Manipulation and DN (Experimental)
  Interventions: Other: HVLA Thrust Manipulation and DN
- Conventional Physical Therapy (Active Comparator)
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: HVLA Thrust Manipulation and DN — HVLA thrust manipulation targeting primarily the lumbar articulations and sacroiliac joint. Up to 10 sessions over 6 weeks. At least one session of dry needling to the lumbo-pelvic muscles and peri-articular ligaments of the SI joint.
  Arms: HVLA Thrust Manipulation and DN
Other: Conventional Physical Therapy — Therapeutic exercise and manual therapy, up to 10 sessions over 6 weeks. Patients may receive interferential current and moist heat.
  Arms: Conventional Physical Therapy

SUMMARY:
The purpose of the research project is to compare the effectiveness of non-thrust mobilization and exercise versus thrust manipulation and dry needling in patients with sacroiliac dysfunction. Physical therapists commonly use both approaches to treat sacroiliac joint dysfunction, and this study is attempting to determine if one approach is more effective than the other.

DETAILED DESCRIPTION:
Patients with sacroiliac pain will be randomized to receive 1-2 treatments per week for 6 weeks (up to 10 sessions total) of either: 1. High-velocity, low-amplitude (HVLA) thrust manipulation and dry needling group, or 2. conventional physical therapy (Stabilization, force closure, motor control exercises and manual therapy) group.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must report sacroiliac dysfunction, defined as:

   * Pain of any duration (acute, subacute, or chronic) in the Fortin region (the pain may also project to the groin, thigh, lower leg and/or foot; however, it may only be local Fortin region pain in some subjects).
   * Pain does NOT centralize with repeated movements or sustained postures
   * A minimum of 3 positive pain provocation tests using either the Laslett et al. (2003, 2005) or van der Wurff et al (2006) multi-test regiments:
   * 3 or more of the following 6 pain provocation tests (Laslett et al, 2003, 2005):
   * Posterior thigh thrust
   * Gaenslen's test (right)
   * Gaenslen's test (left)
   * ASIS distraction
   * ASIS compression
   * Sacral compression
2. A minimum pain rating of 2/10 using the NPRS (Numeric Pain Rating Scale 0---10)
3. A minimum ODI score of 10/50 (i.e. 20% minimum on Oswestry Disability Index)

Exclusion Criteria:

1. Cauda Equina Syndrome
2. Neurologic presentation consistent with upper or lower motor neuron dysfunction due to spinal involvement (ie myelopathy or nerve compression, hyperreflexia, pathologic reflexes, depressed or absent reflexes in the lower extremities, motor weakness involving major muscle groups of lower extremity, unsteady gait, diminished or absent pin prick sensation in the legs and/or feet)
3. Spinal fractures
4. Currently pregnant
5. Co-existing medial problems / comorbidities (e.g., severe osteoporosis, tumors, inflammatory or infectious conditions, diabetes, angina, severe hypertension, RA, etc.)
6. Involvement in litigation of worker's compensation claim for low back
7. Physical therapy or chiropractic treatment for low back pain in the 3 months before initial examination
8. Any indication that might contraindicate spinal manipulative therapy.
9. Recent surgery to the lumbar or thoracic spine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-02-21 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Disability (ODI) | Baseline, 2 Days, 2 Weeks, 6 Weeks, 3 Months
  10 Questions each worth 0-5 points with maximum score of 50 points
Change in Back Pain Intensity (NPRS) | Baseline, 2 Days, 2 Weeks, 6 Weeks, 3 Months
  Numeric Pain Rating
Change in Leg pain Intensity (NPRS) | Baseline, 2 Days, 2 Weeks, 6 Weeks, 3 Months
  Numeric Pain Rating

SECONDARY OUTCOMES:
Change in Medication Intake (Frequency of pain medication) | Baseline, 3 months
  Frequency of pain medication (narcotics and over-the counter drugs) required for low back / pelvic pain

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT FAAOMPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Alabama Physical Therapy & Acupuncture, Montgomery, Alabama, United States